CLINICAL TRIAL: NCT01790373
Title: Suubi+Adherence: Evaluating a Youth-Focused Economic Empowerment Approach to HIV Treatment Adherence
Brief Title: Evaluating a Youth-Focused Economic Empowerment Approach to HIV Treatment Adherence
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Fred Ssewamala, Professor, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: AAAK3852; 1R01HD074949-01 (NIH)
Record Dates: First submitted 2013-02-11; First posted 2013-02-13 (Estimated); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: HIV
Keywords: Suubi; Adolescents; Poverty; Economic empowerment interventions; Adherence to HIV antiretroviral therapy; Wisepill; HIV/AIDS infected Children; Medical event monitoring system; Uganda

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Suubi+Adherence (Experimental): Suubi+Adherence intervention arm provides:
  * Matched savings accounts/child development accounts (CDAs) for the adolescents held in a local bank.
  * Financial education and workshops on asset-building, future planning, and protection from risks
  * Mentorship from a young adult/near-peer
  * Family-based microenterprise development training
  Bolstered Standard of Care: Adherence Counseling Practices
  -Four to six counseling sessions to review HIV, ART, resistance, and adherence.
  Medical Standard of Care:
  -Pediatric ART initiation and monitoring followed by all public clinics, and outlined in National Department of Health Guidelines for pediatric HIV care in Uganda
  Psychosocial Standard of Care:
  -Psychosocial support provided by lay counselors trained in standardized ART adherence counseling
  Interventions: Behavioral: Suubi+Adherence
- Bolstered Standard of Care (Active Comparator): Bolstered Standard of Care: Adherence Counseling Practices
  -Four to six counseling sessions to review HIV, ART, resistance, and adherence.
  Medical Standard of Care:
  -Pediatric ART initiation and monitoring followed by all public clinics, and outlined in National Department of Health Guidelines for pediatric HIV care in Uganda
  Psychosocial Standard of Care:
  -Psychosocial support provided by lay counselors trained in standardized ART adherence counseling
  Interventions: Behavioral: Bolstered Standard of Care

INTERVENTIONS:
Behavioral: Suubi+Adherence — * Matched savings accounts/child development accounts (CDAs) for the adolescents held in a local bank.
  * Financial education and workshops on asset-building, future planning, and protection from risks
  * Mentorship from a young adult/near-peer
  * Family-based microenterprise development training
  * Medical Event Monitoring System
  Bolstered Standard of Care: Adherence Counseling Practices
  -Four to six counseling sessions to review HIV, ART, resistance, and adherence.
  Medical Standard of Care:
  -Pediatric ART initiation and monitoring followed by all public clinics, and outlined in National Department of Health Guidelines for pediatric HIV care in Uganda
  Psychosocial Standard of Care:
  -Psychosocial support provided by lay counselors trained in standardized ART adherence counseling
  Arms: Suubi+Adherence
Behavioral: Bolstered Standard of Care — -Medical Event Monitoring System
  Bolstered Standard of Care: Adherence Counseling Practices
  -Four to six counseling sessions to review HIV, ART, resistance, and adherence.
  Medical Standard of Care:
  -Pediatric ART initiation and monitoring followed by all public clinics, and outlined in National Department of Health Guidelines for pediatric HIV care in Uganda
  Psychosocial Standard of Care:
  -Psychosocial support provided by lay counselors trained in standardized ART adherence counseling
  Arms: Bolstered Standard of Care

SUMMARY:
The goal of Suubi+Adherence is to examine the impact and cost associated with an innovative intervention to increase adherence to HIV treatment for HIV-infected adolescents. Multiple intervention studies by our team in Rakai and Masaka Districts of southern Uganda with AIDS-orphaned adolescents have revealed that if given an opportunity to participate in economic empowerment interventions, youth and their caregivers take full advantage of these interventions to save and invest in their future, show improvements in family financial outcomes, future aspirations, health functioning, sexual-risk taking behaviors, and mental health. The Suubi+Adherence study capitalizes on this prior work, positing that economic empowerment may be a missing, yet critical ingredient to HIV treatment adherence interventions for adolescents and young people. Suubi+Adherence incorporates an economic empowerment design, with a savings-led income generating component, to promote economic stability, and apply it to adherence to HIV treatment regimens for HIV-positive adolescents in a region of southern Uganda with the highest HIV incidence and prevalence in the country.

ELIGIBILITY:
Inclusion Criteria:

* HIV-positive adolescents confirmed by medical report
* Prescribed antiretroviral therapy
* Enrolled in care at one of 40 medical clinics within study region
* 10-16 years of age at the time of enrollment
* Living within a family (not necessarily with biological parent(s))

Exclusion Criteria:

* Not HIV-positive
* HIV-positive but not prescribed antiretroviral therapy
* Not enrolled in care at one of 40 medical clinics within study region
* Younger than 10 years and older than 16 years
* Not living within a family

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 702 (Actual)
Dates: Start 2013-09-07 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline to follow-up assessments of adherence to HIV treatment | Every year for 10 years
  Adherence to HIV treatment regimen outcomes for HIV-positive adolescents, including participants' ability to access and refill prescribed HIV antiretroviral therapy and adhere to prescribed daily HIV medication routines.

SECONDARY OUTCOMES:
Protective Health Behaviors | Every year for 10 years
  Using a series of standardized and pre-tested instruments, potential mechanisms of protective health behaviors, knowledge, and beliefs, including: 1) financial/economic stability, 2) sexual risk-taking behavior, 3) personal beliefs about HIV medication, 4) hopelessness, 5) future plans and aspirations, and 6) adherence self-efficacy, will be measured during a structured interview at baseline and at every subsequent follow-up assessment.
Cost-Effectiveness Analyses | Every year for 10 years
  Cost-effectiveness analyses measure the cost of achieving an agreed upon benefit, such as an additional year of schooling, employment, or a reduction in a disease. Costs will be measured on a per person basis. The costs of the intervention will include all program costs. Research costs will not be included.
Cognitive functioning | Every year in years 6 to 10
  Using a series of standardized and pre-tested instruments, cognitive functioning will be measured during a structured interview at wave 6 and at every subsequent follow-up assessment.
Substance misuse | Every year in years 6 to 10
  Using a series of standardized and pre-tested instruments, substance misuse will be measured during a structured interview at wave 6 and at every subsequent follow-up assessment.
Social transitions | Every year in years 6 to 10
  Using a series of standardized and pre-tested instruments, social transitions will be measured during a structured interview at wave 6 and at every subsequent follow-up assessment.
HIV stigma | Every year in years 6 to 10
  Using a series of standardized and pre-tested instruments, HIV stigma will be measured during a structured interview at wave 6 and at every subsequent follow-up assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Fred M Ssewamala, MSW, PhD, Principal Investigator — Washington University School of Medicine
Locations (2):
- Washington University in St. Louis, St Louis, Missouri, United States
- International Center for Child Health and Asset Development, Masaka, Uganda

REFERENCES:
- [Derived] Tutlam NT, Kizito S, Nabunya P, Naseh M, Nabbosa I, Kwesiga I, Namatovu P, Bahar OS, Nakasujja N, Ssewamala FM. Social Determinants of Mental Health Outcomes Among Refugee Adolescents and Youth Living with HIV in Refugee Settlements in Uganda: A Cross-Sectional Analysis. AIDS Behav. 2025 Nov;29(11):3432-3443. doi: 10.1007/s10461-025-04789-6. Epub 2025 Jun 16. PMID 40518494
- [Derived] Najjuuko C, Brathwaite R, Xu Z, Kizito S, Lu C, Ssewamala FM. Using machine learning to predict poor adherence to antiretroviral therapy among adolescents with HIV in low resource settings. AIDS. 2025 Jul 15;39(9):1204-1213. doi: 10.1097/QAD.0000000000004163. Epub 2025 Feb 24. PMID 39998619
- [Derived] Girma AZ, Brathwaite R, Karamagi Y, Nakabuye F, Nakasujja N, Byansi W, Nabunya P, Sensoy Bahar O, Ssewamala FM. Impact of COVID-19-Related Disruptions on Antiretroviral Therapy Adherence Among Young Adults Living with HIV in Southern Uganda. AIDS Behav. 2025 May;29(5):1640-1649. doi: 10.1007/s10461-025-04634-w. Epub 2025 Feb 10. PMID 39928068
- [Derived] Kizito S, Namuwonge F, Nabayinda J, Nalwanga D, Najjuuko C, Nabunya P, Atwebembere R, Namuyaba OI, Mukasa M, Ssewamala FM. A Cluster-Randomized Controlled Trial of an Economic Strengthening Intervention to Enhance Antiretroviral Therapy Adherence among Adolescents Living with HIV. AIDS Behav. 2024 May;28(5):1570-1580. doi: 10.1007/s10461-024-04268-4. Epub 2024 Jan 17. PMID 38231361
- [Derived] Nabunya P, Samuel K, Ssewamala FM. The effect of family support on self-reported adherence to ART among adolescents perinatally infected with HIV in Uganda: A mediation analysis. J Adolesc. 2023 Jun;95(4):834-843. doi: 10.1002/jad.12157. Epub 2023 Feb 22. PMID 36810778
- [Derived] Kizito S, Namuwonge F, Brathwaite R, Neilands TB, Nabunya P, Bahar OS, Damulira C, Mwebembezi A, Mellins C, McKay MM, Ssewamala FM. Monitoring adherence to antiretroviral therapy among adolescents in Southern Uganda: comparing Wisepill to Self-report in predicting viral suppression in a cluster-randomized trial. J Int AIDS Soc. 2022 Sep;25(9):e25990. doi: 10.1002/jia2.25990. PMID 36052462
- [Derived] Tozan Y, Capasso A, Sun S, Neilands TB, Damulira C, Namuwonge F, Nakigozi G, Mwebembezi A, Mukasa B, Sensoy Bahar O, Nabunya P, Mellins CA, McKay MM, Ssewamala FM. The efficacy and cost-effectiveness of a family-based economic empowerment intervention (Suubi + Adherence) on suppression of HIV viral loads among adolescents living with HIV: results from a Cluster Randomized Controlled Trial in southern Uganda. J Int AIDS Soc. 2021 Jun;24(6):e25752. doi: 10.1002/jia2.25752. PMID 34176245
- [Derived] Ssewamala FM, Sensoy Bahar O, Nabunya P, Thames AD, Neilands TB, Damulira C, Mukasa B, Brathwaite R, Mellins C, Santelli J, Brown D, Guo S, Namatovu P, Kiyingi J, Namuwonge F, McKay MM. Suubi+Adherence-Round 2: A study protocol to examine the longitudinal HIV treatment adherence among youth living with HIV transitioning into young adulthood in Southern Uganda. BMC Public Health. 2021 Jan 21;21(1):179. doi: 10.1186/s12889-021-10202-3. PMID 33478469
- [Derived] Nabunya P, Bahar OS, Chen B, Dvalishvili D, Damulira C, Ssewamala FM. The role of family factors in antiretroviral therapy (ART) adherence self-efficacy among HIV-infected adolescents in southern Uganda. BMC Public Health. 2020 Mar 17;20(1):340. doi: 10.1186/s12889-020-8361-1. PMID 32183762
- [Derived] Ssewamala FM, Dvalishvili D, Mellins CA, Geng EH, Makumbi F, Neilands TB, McKay M, Damulira C, Nabunya P, Sensoy Bahar O, Nakigozi G, Kigozi G, Byansi W, Mukasa M, Namuwonge F. The long-term effects of a family based economic empowerment intervention (Suubi+Adherence) on suppression of HIV viral loads among adolescents living with HIV in southern Uganda: Findings from 5-year cluster randomized trial. PLoS One. 2020 Feb 10;15(2):e0228370. doi: 10.1371/journal.pone.0228370. eCollection 2020. PMID 32040523
- [Derived] Ssewamala FM, Byansi W, Bahar OS, Nabunya P, Neilands TB, Mellins C, McKay M, Namuwonge F, Mukasa M, Makumbi FE, Nakigozi G. Suubi+Adherence study protocol: A family economic empowerment intervention addressing HIV treatment adherence for perinatally infected adolescents. Contemp Clin Trials Commun. 2019 Oct 20;16:100463. doi: 10.1016/j.conctc.2019.100463. eCollection 2019 Dec. PMID 31872152